CLINICAL TRIAL: NCT00525954
Title: Phospholipase Levels And Serological Markers of Atherosclerosis 2: An Examination of Once Daily (QD) Dosing of A-002 In Subjects With Stable Coronary Artery Disease
Brief Title: PLASMA 2 Trial: Examination of Once Daily (QD) Dosing of A-002 In Subjects With Stable Coronary Artery Disease
Acronym: PLASMA 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anthera Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AN-CVD2222
Record Dates: First submitted 2007-09-04; First posted 2007-09-06 (Estimated); Last update posted 2008-01-07 (Estimated); Status verified 2008-01

CONDITIONS: Coronary Artery Disease
Keywords: Coronary; Artery; Artheroschlerosis; Phospholipase; CAD; Coronary Artery Disease (CAD)
MeSH Terms: conditions — Coronary Artery Disease | interventions — varespladib methyl

INTERVENTIONS:
Drug: A-002

SUMMARY:
The study will be conducted at up to 25 U.S. centers and will be a double-blind randomized parallel group placebo controlled study among subjects with stable coronary artery disease (CAD). Subjects will be randomized to receive either placebo tablets or one of 2 orally active doses of A-002. The duration of study drug therapy will be 8 weeks.

DETAILED DESCRIPTION:
A-002 represents a novel therapy for the treatment of atherosclerosis and coronary artery disease (CAD). Through the inhibition of activity A-002 may provide multifunctional activity directed against key facets of the disease process, namely a) inflammation, b) atherogenic lipid profiles and c) the atherosclerotic process. Non-clinical and clinical data from recent studies have demonstrated the benefit of early and aggressive anti-inflammatory therapy to reduce cardiovascular risk. Recent clinical studies have provided a strong association between levels and cardiovascular event risk. The proposed Phase 2 clinical pharmacology study (Study No. AN-CVD-2222) will examine the effects of 2 different doses of A-002 compared with placebo, on enzyme levels and activity after 8 weeks of treatment. In addition, the effect of treatment on inflammatory markers of cardiovascular risk (C-reactive protein [CRP]), lipid levels and lipoprotein subclasses and other soluble biomarkers (e.g., ICAM-1, VCAM-1, TNF, MCP-1 etc) will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible for inclusion if they meet the following inclusion criteria:

1. Men and women ≥18 years of age
2. Written informed consent from the subject
3. Stable CAD
4. Stable medical condition, will be compliant and able to comply with the requirements of the protocol

Exclusion Criteria:

Subjects must NOT meet any of the following exclusion criteria:

1. Planned coronary artery bypass surgery (CABG)
2. Acute or chronic heart failure as defined by the New York Heart Association (NYHA) classification as functional Class III or Class IV
3. Hospitalization for acute coronary syndrome (ACS) if troponin >0.1 ng/mL in the preceding 6 weeks
4. Hospitalization for ST-segment elevation acute myocardial infarction (STEMI) in the preceding 12 weeks
5. Subjects with chronic inflammatory disease (e.g., rheumatoid arthritis), inflammatory bowel disease, recent (12 weeks) systemic or localized infection (the latter requiring clinical intervention), or major surgery
6. hs-CRP ≥15 mg/L repeated on at least 2 occasions >24 hours apart due to non-cardiovascular systemic inflammatory conditions (e.g., rheumatoid disease)
7. Subjects enrolled in another experimental (interventional) protocol within the past 30 days prior to Screening or prior experience with A-002.
8. Subjects treated for cancer within the previous 5 years except for skin basal cell carcinoma or carcinoma in situ of the cervix, with measures other than a minor, complete surgical excision (e.g., chemotherapy), or radiation therapy
9. Subjects who have received immunosuppressant therapy within 30 days prior to entry
10. Subjects who have received anti-tumor necrosis factor (for example, infliximab) therapy within 6 months prior to entry
11. The presence of severe liver disease with cirrhosis, recent active hepatitis, active chronic hepatitis, ALT or AST >3 x upper limit of normal, biliary obstruction with hyperbilirubinemia (total bilirubin >2 x upper limit of normal)
12. Active cholecystitis, gall bladder symptoms, or potential hepato-biliary abnormalities
13. The presence of moderate or severe renal impairment (CrCl <60 mL/min or creatinine >1.5 x upper limit of normal), nephrotic syndrome, or subjects undergoing dialysis
14. Uncontrolled diabetes mellitus (known HbA1c >11% within the last 1 month prior to screening)
15. Females who are nursing, pregnant, or intend to become pregnant during the time of the study, or subjects who have a positive serum pregnancy test at Visit 1 (if the subject is a female of child-bearing potential). Women of child-bearing potential must also use a reliable method of birth control during the study and for 1 month following completion of therapy. A reliable method for this study is defined as one of the following: oral or injectable contraceptives, intrauterine device (IUD), contraceptive implants, tubal ligation, hysterectomy, a double-barrier method (diaphragm with spermicidal foam or jelly, or a condom).
16. Subjects who have a history of alcohol or drug abuse within 1 year of study entry
17. Subject living too far from participating center or unable to return for follow-up visits
18. Subjects who in the opinion of the Investigator are a poor medical or psychiatric risk for therapy with an investigational drug, are unreliable, or have an incomplete understanding of the study which may affect their ability to take drugs as prescribed or comply with instructions
19. Known human immunodeficiency virus (HIV), Hepatitis B virus (HBV), or Hepatitis C Virus (HCV) infection
20. Treatment with any systemic corticosteroid within the 30-day period prior to study entry or the use of inhaled steroids within the 14-day period prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2007-09; Study Completion 2007-12

PRIMARY OUTCOMES:
The primary objective of this study is to determine the effect of once daily (QD) dosing of A-002 on sPLA2 levels and activity

SECONDARY OUTCOMES:
Determine the effect of QD dosing of A-002 on sPLA2 levels and activity at each time point (Weeks 2, 4, and 8)
Compare the effect of QD dosing of A-002 on sPLA2 enzyme levels and markers of inflammation
Determine plasma drug concentrations with QD dosing

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Mobile Heart Specialists, Mobile, Alabama
  - Sonoran Health Specialists, Scottsdale, Arizona
  - Pasco Cardiology Center, Hudson, Florida
  - Charlotte Cardiovascular Institute, Port Charlotte, Florida
  - Florida Cardiovascular Research Institute, Tampa, Florida
  - Augusta Cardiology Clinic, Augusta, Georgia
  - Louisville Cardiology Medical Group, Louisville, Kentucky
  - Maine Research Associates, Auburn, Maine
  - United Medical Associates, Binghamton, New York
  - Cardiology PC, Syracuse, New York
  - Austin Heart, Austin, Texas
  - Clinical Research Associates of Tidewater, Norfolk, Virginia
  - Wisconsin Heart, SC, Madison, Wisconsin

REFERENCES:
- [Derived] Rosenson RS, Elliott M, Stasiv Y, Hislop C; PLASMA II Investigators. Randomized trial of an inhibitor of secretory phospholipase A2 on atherogenic lipoprotein subclasses in statin-treated patients with coronary heart disease. Eur Heart J. 2011 Apr;32(8):999-1005. doi: 10.1093/eurheartj/ehq374. Epub 2010 Nov 16. PMID 21081550